CLINICAL TRIAL: NCT03033225
Title: Phase II Study of EUS-Guided Verteporfin PDT in Solid Pancreatic Tumors (VERTPAC-02)
Brief Title: Ultrasound-Guided Verteporfin Photodynamic Therapy for the Treatment of Unresectable Solid Pancreatic Tumors or Advanced Pancreatic Cancer, VERTPAC-02 Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-001243; NCI-2019-07003 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16-001243 (Other: Mayo Clinic in Rochester); P01CA084203 (NIH)
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2023-12

CONDITIONS: Advanced Pancreatic Carcinoma; Locally Advanced Pancreatic Carcinoma; Metastatic Pancreatic Carcinoma; Pancreatic Neoplasm; Stage II Pancreatic Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Unresectable Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration; Optical Imaging; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Phototherapy; Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (verteporfin, EUS-guided PDT) (Experimental): Patients receive verteporfin IV and undergo fluorescence imaging and after 60 minutes undergo EUS-guided PDT.
  Interventions: Procedure: Endoscopic Ultrasound; Procedure: Fluorescence Imaging; Drug: Photodynamic Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Verteporfin

INTERVENTIONS:
Procedure: Endoscopic Ultrasound — Undergo EUS-guided PDT
  Other Names: endosonography; EUS
Procedure: Fluorescence Imaging — Undergo fluorescence imaging
Drug: Photodynamic Therapy — Undergo EUS-guided PDT
  Other Names: PDT; Photoradiation Therapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Verteporfin — Given IV
  Other Names: Benzoporphyrin Derivative Monoacid Ring A; BPD-MA; Visudyne

SUMMARY:
This phase II trial studies how well ultrasound-guided verteporfin photodynamic therapy works for the treatment of patients with solid pancreatic tumors that cannot be removed by surgery (unresectable) or pancreatic cancer that has spread to other places in the body (advanced). Photodynamic therapy is a type of laser device that is guided by ultrasound imaging and used in combination with the drug verteporfin that may be less invasive and as effective as current treatment methods for patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To show that endoscopic ultrasound (EUS)-guided photodynamic therapy (PDT) to the pancreas is effective at direct ablation of advanced or locally advanced and small volume metastatic pancreatic tumors in a multicenter setting.

SECONDARY OBJECTIVE:

I. To evaluate the predictability of tumor necrosis as a function of delivered energy, based on pre-PDT contrast computed tomography (CT) scans.

TERTIARY OBJECTIVE:

I. Evaluate the safety of chemotherapy given two days after PDT.

QUARTERNARY OBJECTIVE:

I. Demonstrate that cancer biomarkers in pre- versus (vs.) post-PDT are surrogate markers of response.

OUTLINE:

Patients receive verteporfin intravenously (IV) and undergo fluorescence imaging and after 60 minutes undergo EUS-guided PDT.

After completion of study treatment, patients are followed up at 14 days, and at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological diagnosis (Dx) of advanced or locally advanced or small volume metastatic pancreatic cancer (PanCa) or other solid pancreatic tumor that is not amenable to curative surgical resection, or the patient is unfit, or declines surgery
* Age > 18 years
* Measurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST)
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Estimated life expectancy of at least 12 weeks
* Capable of giving written informed consent
* Adequate biliary drainage (serum bilirubin < 2.5 upper limit of normal [ULN]), with no evidence of active uncontrolled infection (patients on antibiotics are eligible)
* Women of child-bearing potential with a negative pregnancy test (qualitative serum human chorionic gonadotropin [HCG]) prior to study entry AND must be using an adequate contraception method, which must be continued for 1 week after PDT

Exclusion Criteria:

* For locally advanced patients, evidence of metastases other than lung or liver. For lung metastases, greater than three lesions and any lesions greater than 5 cm are excluded. For advanced patients, any metastasis is acceptable for enrollment
* Porphyria
* Pregnant or breast-feeding
* Locally advanced disease involving > 50% circumference of the duodenum or a major artery within the treatment area
* ECOG performance status 3 or 4
* Previous treatment with curative intent for current disease within the past two weeks (i.e. prior resection, radical radiotherapy or chemotherapy)
* Any psychiatric disorder making reliable informed consent impossible
* A history of documented hemorrhagic diathesis or coagulopathy on therapeutic anticoagulation
* History of prior or concomitant other malignancy that will interfere with the response evaluation
* Any evidence of severe or uncontrolled systemic diseases or laboratory finding that in the view of the investigator makes it undesirable for the patient to participate in the trial
* Contrast allergy not amenable to treatment with steroids and antihistamines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Chandrasekhara, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Hanada Y, Pereira SP, Pogue B, Maytin EV, Hasan T, Linn B, Mangels-Dick T, Wang KK. EUS-guided verteporfin photodynamic therapy for pancreatic cancer. Gastrointest Endosc. 2021 Jul;94(1):179-186. doi: 10.1016/j.gie.2021.02.027. Epub 2021 Feb 26. PMID 33647286
- [Derived] Vincent P, Maeder ME, Hunt B, Linn B, Mangels-Dick T, Hasan T, Wang KK, Pogue BW. CT radiomic features of photodynamic priming in clinical pancreatic adenocarcinoma treatment. Phys Med Biol. 2021 Aug 23;66(17):10.1088/1361-6560/ac1458. doi: 10.1088/1361-6560/ac1458. PMID 34261044
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 15, 2017 and July 20, 2019, 623 potential patients were examined for eligibility. Of these, 54 were confirmed eligible and approached for consideration. Eight participants proceeded to inclusion/study completion. Reasons for nonparticipation included nonresponse, unsuitable timing of study (for personal reasons or decision to initiate a chemotherapeutic agent), unsuitable location of study/unwillingness to travel to study site, and entry into a different research study.
Groups:
- Treatment (Verteporfin, EUS-guided PDT): Patients receive verteporfin IV and undergo fluorescence imaging and after 60 minutes undergo Endoscopic Ultrasound (EUS)-guided Photodynamic therapy (PDT).
Period: Overall Study
Arm/Group | Treatment (Verteporfin, EUS-guided PDT)
Started | 13
Completed | 8
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Verteporfin, EUS-guided PDT)
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Assessed by the number of participants who did or did not respond, evaluated by tumor necrosis as a function of delivered energy, based on pre-photodynamic therapy (PDT) contrast computed tomography (CT) scans. Tumor volume response was graded per Response Evaluation Criteria in Solid Tumors (RECIST) criteria. CT scans were obtained on day 2 following PDT. Most patients (87.5%) had a repeat CT of the abdomen and pelvis for reasons unrelated to the study; these CTs were also reviewed for tumor response.
Time Frame: Baseline (up to 28 days before PDF); 2 days post PDT; Up to 12 months post PDT
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Verteporfin, EUS-guided PDT)
Number analyzed (Participants) | 8
Participants
  PDT Response | 5
  PDT Non-response | 3

ADVERSE EVENTS:
Time Frame: Adverse event monitoring occurring on days 1, 2, and 14 following PDT.
Arm/Group | Treatment (Verteporfin, EUS-guided PDT)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT03033225/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT03033225/ICF_001.pdf